CLINICAL TRIAL: NCT05536752
Title: A Phase 2, Double-Masked, Randomized, Placebo-Controlled, Dose-Response Study Assessing the Safety and Efficacy of QA102 in Subjects With Dry Age-Related Macular Degeneration (AMD)
Brief Title: QA102 Phase II Study in Subjects With Dry AMD
Acronym: AMEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Smilebiotek Zhuhai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QA102-CS201
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Dry Age-related Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- QA102 200mg group (Experimental): Subjects randomized to this arm will receive one (1) 200 mg capsule of QA102 and 1 placebo capsule BID = daily dose of 400 mg QA102 for up to 15 months
  Interventions: Drug: QA102/Placebo
- QA102 400mg group (Experimental): Subjects randomized to this arm will receive two (2) 200 mg capsules of QA102 BID = daily dose of 800 mg QA102 for up to 15 months
  Interventions: Drug: QA102
- Placebo group (Placebo Comparator): Subjects randomized to this arm will receive two (2) placebo capsules BID = daily dose of 0 mg QA102 for up to 15 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QA102/Placebo — Capsules
  Arms: QA102 200mg group
Drug: QA102 — Capsules
  Arms: QA102 400mg group
Drug: Placebo — Capsules
  Arms: Placebo group

SUMMARY:
This is a phase 2, double-masked, randomized, placebo-controlled, dose-response study. The primary objective of the study is to evaluate the efficacy of QA102 oral capsules on the development of soft drusen, visual acuity (VA), and geographic atrophy (GA) or choroidal neovascularization (CNV) or the progression of GA in subjects with intermediate to advanced dry AMD.

DETAILED DESCRIPTION:
Approximately 30 sites will randomize a total of approximately 150 subjects to 1 of 3 treatment arms in a 1:1:1 ratio (50 subjects per arm). Each subject will receive either QA102 or matching placebo BID for up to 15 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject must be able to understand and willing to sign a written informed consent form (ICF) prior to the initiation of any study-specific procedures.
* Subject must be age ≥50 years at the time of informed consent.
* Subject must be able to take oral medications and willing to record daily adherence to taking their assigned capsules.
* Subject must have adequate hematologic function, hepatic function, renal function and coagulation profile as defined in the protocol.
* Subject must be willing and able to comply with study procedures and examinations.

Specific to the Study Eye:

* Subject must have one of the following:

  * extensive intermediate-size drusen, or at least 1 large drusen, or
  * GA ((not involving the foveal center point) secondary to AMD, with very limited aggregate size of total GA(s), as defined in the protocol.
* Subject must be able to correctly identify ≥35 ETDRS letters (approximately 20/200 Snellen equivalent).

Specific to Fellow Eye:

- Subject must have a diagnosis of advanced AMD (evidence of GA and/or CNV), to be confirmed by the CRC.

Specific to Both Eyes:

- Subject must have visualizable retina, clear ocular media, and adequate pupillary dilation to ensure high-quality fundus imaging.

Key Exclusion Criteria:

* Subject received an active investigational drug within 6 weeks (or 5 half-lives of the active, whichever is longer) prior to screening for this QA102 study.
* Subject has ever received gene therapy (for any condition).
* Subject is unwilling to stop intake of Age-Related Eye Disease Studies (AREDS) vitamins for the duration of the study.
* Subject has a clinically significant systemic disease that might interfere with the study, in the judgment of the Investigator.
* Subject had major surgery within 30 days prior to Screening.

Specific to Study Eye:

* Subject has large GA, subfoveal GA, or active or inactive CNV, as confirmed by the CRC.
* Subject has GA or CNV due to causes other than AMD that that developed between Visit 1 (Screening) and Visit 2 (Randomization).
* Subject has endophthalmitis.
* Subject has a hemorrhagic or serous pigment epithelial detachment (PED) within 500 µm of the foveal center point, to be confirmed by the CRC.
* Subject has had retinal procedures or surgeries, or has a retinal pathology, such as a macular hole.
* Subject has aphakia or absence of the posterior capsule.
* Subject has ever received, whether in an interventional trial or by prescription, an FDA- approved treatment for GA. Use of such treatment during the QA102 study period also is prohibited. (Study Eye Only)

Specific to Fellow Eye:

Subject has monocular vision impairment, defined as having no light perception in the fellow eye with adequate vision in the study eye.

Specific to Either Eye:

* Subject had intraocular surgery with lens replacement within 3 months of Screening.
* Subject has any ophthalmic condition that could require surgery during the study period.
* Subject has an ocular condition that might affect adequate imaging of the retina and/or or alter visual acuity.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in soft drusen volume (mm3) | Month 12
  In the study eye at Month 12, change from baseline in best-corrected visual acuity (BCVA) as measured by Early Treatment Diabetic Retinopathy Study (ETDRS).

SECONDARY OUTCOMES:
Change from Baseline in BCVA | Month 12
  Change from Baseline in best-corrected visual acuity (BCVA) at month 12 as measured by Early Treatment Diabetic Retinopathy Study (ETDRS).
Change from Baseline in LLVA | Month 12
  In the study eye at Month 12, change from baseline in low-luminance visual acuity (LLVA) as measured by ETDRS.
Change from baseline in soft drusen volume (mm3) | Month 1,2,3,6,9,12,15
  Change from baseline in drusen volume (mm3) as measured by SD-OCT at time points other than Month 12 (study eye) or at all time points (fellow eye).
Change from Baseline in BCVA | Month 1,2,3,6,9,12,15
  Change from baseline in BCVA as measured by ETDRS at time points other than Month 12 (study eye) or at all time points (fellow eye).
Change from Baseline in LLVA | Month 1,2,3,6,9,12,15
  Change from baseline in LLVA as measured by ETDRS at time points other than Month 12 (study eye) or at all time points (fellow eye).
Change from baseline in GA | Month 1,2,3,6,9,12,15
  Change from baseline in GA area as measured by fundus autofluorescence (FAF) and/or SD-OCT.
Change from baseline in GA | Month 1,2,3,6,9,12,15
  Change from baseline in GA area as measured by the square root transformation of area on FAF and/or SD-OCT.
Mean rate of GA growth | Month 1,2,3,6,9,12,15
  In the study eye, the estimated mean rate of growth (slope) based on GA area measured by FAF at ≥3 time points.
Area under the curve for BCVA letters | Month 1,2,3,6,9,12,15
  Area under the curve for BCVA letters read on the ETDRS chart over the 15-month treatment period.
Proportion of subjects with disease progression | Month 15
  In the study eye at Month 15, proportion of subjects with disease progression, defined as (a) development of CNV, as assessed by SD-OCT and/or FAF, or (b) GA change from baseline of ≥0.50 mm2, as assessed by FAF. Both assessments will be conducted by the central reading center (CRC).
Proportion of subjects with progression of GA | Month 1,2,3,6,9,12,15
  Proportion of subjects with progression of GA, defined as a change from baseline of ≥0.50 mm2, at time points other than Month 15 (study eye) or at all time points (fellow eye), as determined by the CRC using FAF and/or SD-OCT.
Rescue injections | Month 1,2,3,6,9,12,15
  Proportion of subjects requiring rescue injections of anti-VEGF therapies for CNV.
iRORA | Month 1,2,3,6,9,12,15
  Proportion of subjects developing new incomplete retinal pigment epithelium and outer retinal atrophy (iRORA), as determined by the CRC.
Fellow eye CNV | Month 1,2,3,6,9,12,15
  Proportion of subjects with CNV achieving optimal control of CNV, defined as the absence of subretinal fluid (SRF), at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Retina Associates - Plano, Plano, Texas, United States